CLINICAL TRIAL: NCT00329563
Title: Pilot Community Clinical Study of Hypothermia in Cardiac Arrest
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Medic One Foundation (Other)
Responsible Party: Principal Investigator, Francis Kim, Associate Professor, Medicine, Division of Cardiology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25186
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest; Hypothermia
MeSH Terms: conditions — Heart Arrest; Hypothermia

ARMS (2):
- Cold fluid (Experimental)
  Interventions: Drug: Up to 2 liter infusion of cold 4 degree C normal saline
- control, standard of care (No Intervention)

INTERVENTIONS:
Drug: Up to 2 liter infusion of cold 4 degree C normal saline — Patients randomized to field cooling will receive up to 2 liters of 4oC normal saline. Control patients will receive standard of care following resuscitation.
  Arms: Cold fluid

SUMMARY:
The overall goal of this study is to determine the feasibility of initiating hypothermia in cardiac arrest patients as soon as possible in the field. In this pilot study we will randomize 125 patients after return of spontaneous circulation (ROSC) to hypothermia with rapid infusion of 2 liters of 4oC Normal Saline IV solution over 20 to 30 minutes, IV sedation and muscle paralysis or to standard of care following ROSC. The primary objectives of this study will be to determine whether temperature of 33-34oC can be achieved and maintained using this strategy. The primary outcome measures will include: temperature changes of the patients at time of admission to the hospital. Secondary analysis will include determining if the proportion of patients discharged from the hospital is increased in the group receiving hypothermia. If this initial pilot study can demonstrate feasibility in achieving and maintaining hypothermia, a larger randomized clinical trial to test the hypothesis that hypothermia initiation in the field will increase the proportion of patients surviving following cardiac arrest will be planned.

ELIGIBILITY:
Inclusion Criteria:

* Resuscitated out-of-hospital cardiac arrest defined as having a palpable pulse comatose IV access Intubated

Exclusion Criteria:

* age less than 18 traumatic cause of cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2004-11; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Temperature difference between first field temperature and hospital arrival temperature | less than 60 minutes

SECONDARY OUTCOMES:
Survival to discharge from hospital | Between 2 -30 days
Awakening in the hospital | between 2-30 days

CONTACTS AND LOCATIONS:
Overall Officials: Francis Kim, MD, Principal Investigator — University of Washington